CLINICAL TRIAL: NCT03995121
Title: Synaptic Density in Psychiatric Disorders Using SV2A Receptor PET Imaging With [11C]APP311
Brief Title: SV2 PET Imaging With [11C]APP311
Acronym: SV2
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Other Study IDs: 2000021592; 1R01DA054314-01 (NIH); 36C24820C0079 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia and Other Psychotic Disorders; Cannabis Use Disorder; Healthy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — When specimens and information are stored, researchers are careful to try to protect your identity from discovery by others. Samples and information will receive a unique code. Other researchers will only receive coded samples and information, and will not be able to link the code to subjects. Strict security safeguards are in place to reduce the chance of misuse or unplanned release of information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Schizophrenia and other psychotic disorders: For each [11C]APP311 PET scan, up to 20 mCi of [11C]APP311 will be administered by infusion pump, followed by up to 120 minutes of dynamic PET data acquisition.
  Interventions: Drug: [11C]APP311
- Cannabis Use Disorder: For each [11C]APP311 PET scan, up to 20 mCi of [11C]APP311 will be administered by infusion pump, followed by up to 120 minutes of dynamic PET data acquisition.
  Interventions: Drug: [11C]APP311
- Healthy Control: For each [11C]APP311 PET scan, up to 20 mCi of [11C]APP311 will be administered by infusion pump, followed by up to 120 minutes of dynamic PET data acquisition.
  Interventions: Drug: [11C]APP311

INTERVENTIONS:
Drug: [11C]APP311 — It has been shown that radiotracer [11C]APP311 (aka [11C]UCB-J) displays high specificity and selectivity for the synaptic vesicle protein SV2A. Since this protein is expressed ubiquitously in active synapses, this tracer has the potential to be a general purpose tool for quantitative imaging of synaptic density.

SUMMARY:
The aim of this study is to evaluate a new SV2A tracer, [11C]APP311, in healthy aging and neuropsychiatric disorders including psychotic disorders and cannabis use disorders.

DETAILED DESCRIPTION:
The overall goal of this protocol is to study synaptic density in two psychiatric disorders (namely schizophrenia and other psychotic disorders, and cannabis use disorder) with this exciting new PET tracer. Secondary outcomes will include electroencephalography (EEG). A battery of EEG paradigms assessing sensory, perceptual, and cognitive functions will also be administered. The primary dependent measures will be traditional event related potentials (ERPs; e.g. latency and amplitude) as well as time X frequency analysis (inter-trial coherence and spectral power).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give voluntary written informed consent
* Male and Female subjects, age 18 to 65 years, inclusive

Exclusion Criteria:

* MRI metal exclusions and claustrophobia.
* Education completed is less than 12 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruiting Subjects with Schizophrenia and other Psychotic disorders Cannabis Use Disorder Healthy controls
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Synaptic density in psychiatric disorders using SV2A receptor PET Imaging with [11C]APP311 | One test day (one time point).
  To compare synaptic vesicle protein 2A (SV2A) density in two groups of subjects with psychiatric disorders (namely 'schizophrenia and other psychotic disorders', and 'cannabis use disorder') to that in healthy controls using the PET radiotracer 11C-APP311

SECONDARY OUTCOMES:
Correlation of Synaptic density with cognition and EEG | One test day (one time point).
  To correlate SV2A density with concurrent measures of information processing such as cognitive performance on a neuropsychiatric battery and electroencephalographic (EEG) measures

CONTACTS AND LOCATIONS:
Locations (1):
- Conneticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No